CLINICAL TRIAL: NCT05112991
Title: An Open-label, Multi-center, Multi-corhort Phase II Study of Envafolimab Alone or With Lenvatinib in Patients With Advanced Endometrial Cancer
Brief Title: Study of Envafolimab Alone or With Lenvatinib in Patients With Advanced Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KN035-CN-011
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced Endometrial Cancer
Keywords: endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — envafolimab

STUDY DESIGN:
Intervention Model Description: This study is an open-label, two-arm study, without randomization and blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envafolimab + Lenvatinib (Experimental): Subjects receive lenvatinib daily and envafolimab once on Day 1 and 15 of the first cycle and at the beginning of each subsequent 4 week treatment cycle D1.
  Interventions: Drug: Envafolimab+Lenvatinib
- Envafolimab (Experimental): Subjects receive envafolimab once on Day 1 and 15 of the first cycle and at the beginning of each subsequent 4 week treatment cycle D1.
  Interventions: Drug: Envafolimab

INTERVENTIONS:
Drug: Envafolimab+Lenvatinib — Envafolimab: 400mg envafolimab was administered once in D1 and D15 of the first treatment cycle and once in D1 of each subsequent 28 day cycle.
  Lenvatinib: the recommended Phase 2 dose (RP2D) orally 20mg QD during each 28-day cycle.
  Arms: Envafolimab + Lenvatinib
Drug: Envafolimab — Envafolimab: 400mg envafolimab was administered once in D1 and D15 of the first treatment cycle and once in D1 of each subsequent 28 day cycle.
  Arms: Envafolimab

SUMMARY:
This is an open-label, multi-center, multi-corhort Phase II study of Envafolimab alone or with Lenvatinib in patients with advanced endometrial cancer.The primary objective is to evaluate objective response rate of envafolimab alone or with lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent form.
2. Has a histologically confirmed diagnosis of endometrial carcinoma (EC). Has Documented evidence of advanced, recurrent or metastatic EC and are not candidates for curative surgery or radiation.
3. Failure or intolerance of standard first-line platinum-based chemotherapy regimen for EC.

   Note: If recurrence occurs during adjuvant/neoadjuvant therapy or within 12 months after completion, adjuvant/neoadjuvant therapy is considered to be the first-line treatment for advanced disease. There is no restriction regarding prior hormonal therapy.
4. Has at least 1 measurable target lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and confirmed by Blind Independent Imaging Review Committee (BIRC).
5. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of 12 weeks or more.
7. Sufficient organ and bone marrow function (no hematopoietic growth factor, blood transfusion or platelet therapy was given within 14 days before the first study drug treatment).
8. Archival tumor tissue or a newly obtained biopsy must be available prior to the first dose of study drug for biomarker analysis. Tissue samples need to be from lesions that have not received local radiotherapy.
9. Females of childbearing potential must have a negative serum pregnancy test within 7 days of the first dose of study drug.

Exclusion Criteria:

1. Previous lab results showed dMMR or MSI-H.
2. Participate in the clinical trials of other investigational drugs within 28 days before the first medication; or have received anti-tumor treatment within 2 weeks, including but not limited to chemotherapy and radiotherapy or targeted therapy.
3. The toxicity of previous anti-tumor treatments has not recovered to 0 or 1 level.
4. Recieved major surgery with 28 days before the first medication or has serious nonhealing wound, ulcer, or bone fracture at screening.
5. Has received prior treatment with any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
6. Uncontrolled blood pressure (BP) with or without antihypertensive medications, defined as BP >150/90 mmHg.
7. Uncontrolled or major Cardio-cerebral vascular disease.
8. Have active, or have had autoimmune diseases or risks that may recur. However, subjects required only replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) or with skin diseases that do not require systemic treatmentare are allowed to be included.
9. Subjects who need to use corticosteroids (> 10 mg/day prednisone equivalent dose) for systemic therapy within 14 days before the study drug is administered.
10. Has received a live-virus vaccination within 28 days of planned treatment start or plan to reveived a live-virus vaccination during the study.
11. Has current or suspected (non-infectious) pneumonitis.
12. Active infection (any infection requiring systemic treatment).
13. Has active Hepatitis B or C.
14. Is positive for Human Immunodeficiency Virus (HIV).
15. Has uncontrolled pericardial effusion, pleural effusion or ascites.
16. Has symptomatic/active brain metastasis or meningeal carcinomatosis; for patients with brain metastases who have previously received treatment, if the clinical and imaging evidence does not indicate disease progression within 4 weeks before the first study drug treatment, and 2 weeks before the first administration There is no need to receive corticosteroid treatment and can be considered for inclusion.
17. Suffered from other known malignant tumors within 5 years before enrollment (except for treated skin basal cell carcinoma, skin squamous cell carcinoma and/or carcinoma in situ after radical resection).
18. Hypersensitivity to either of the study drug or its components.
19. Females who are pregnant or breastfeeding and who refuse to use a highly effective method of contraception throughout the entire study period, and for 6 months after the last dose of study drug;
20. According to the judgement of the investigators, there are other factors indicate that the subject should not be enrolled.
21. Has received prior treatment with any treatment targeting VEGF-directed angiogenesis.
22. Has radiographic evidence of major blood vessel invasion/infiltration.
23. Has a history of hypertensive crisis or hypertensive encephalopathy.
24. Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
25. Has a history of serious bleeding disease within 6 months prior to the first dose of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR of Envafolimab alone or with Lenvatinib | Up to approximately 24 months
  The ORR (either confirmed complete response [CR] or partial response [PR]) based on RECIST 1.1 will be determined in participants who have measurable disease at study entry.

SECONDARY OUTCOMES:
The duration of response (DoR） | Up to approximately 24 months
Disease control rate (DCR) | Up to approximately 24 months
Time to response (TTR) | Up to approximately 24 months
Progression-free survival (PFS) | Up to approximately 24 months
To evaluate the overall survival (OS) in in subjects with advance endometrial cancer | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: xiaohua Wu, Dr, Principal Investigator — Fudan University
Locations (19):
- China (19):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - :Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Yueyang Center Hospital, Yueyang, Hunan
  - :Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - :Linyi Cancer Hospital, Linyi, Shandong
  - Tai'an Center Hospital, Tai’an, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute&Hospital, Tianjing, Tianjing
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No